CLINICAL TRIAL: NCT04541992
Title: Body-Worn Sensors for Risk of Injury Prediction During Military Training
Brief Title: Sensors Prediction Study
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: The Geneva Foundation (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Gailey, Professor, University of Miami
Other Study IDs: 20190910; HU00011920011 (Other Grant/Funding Number: Geneva Foundation)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Injury Leg
Keywords: hip injury; knee injury; ankle injury
MeSH Terms: conditions — Leg Injuries; Hip Injuries; Knee Injuries; Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Airborne Group: Participants in this group will be tested for balance and agility within a 20 minute time frame.

SUMMARY:
The purpose of this study is to test whether measures of balance and agility can help predict if a Service Member may be at risk for an injury to their legs before beginning their school and training.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-55
2. Active duty Service Members in the 82nd Airborne Division (ABN DIV)
3. Fluent in English speak and reading

Exclusion Criteria:

1. Service members under the age of 18 or over the age of 55 will be excluded
2. Told by a doctor that they should not exercise.
3. Orthopedic injury/surgery of the lower limb or back within the last year and that limits study compliance
4. Regular use of medications that may alter balance, coordination or agility
5. Unwilling to comply with the study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy service member participants stationed at Fort Bragg, North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 8300 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Region of Limb Stability | Day 1
  Region of Limb Stability (ROLS) measured in cm^2 using a body-worn sensor.
Transitional Angular Displacement of Segments | Day 1
  Transitional Angular Displacement of Segments (TADS) measured in degrees per second using a body-worn sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gailey, PhD, Principal Investigator — University of Miami
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No